CLINICAL TRIAL: NCT04195919
Title: A Clinical Study to Investigate the Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of Evogliptin in Hemodialysis Patients
Brief Title: The Pharmacokinetics/Pharmacodynamics and Safety/Tolerability of Evogliptin in Hemodialysis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DA1229_ESRD_I
Record Dates: First submitted 2019-12-04; First posted 2019-12-12 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Hemodialysis Patients
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): Hemodialysis patients(MDRD-eGFR ≤ 15 mL/min/1.73m2)
  Interventions: Drug: Evogliptin 5mg
- Group2 (Experimental): Healthy control(MDRD-eGFR ≥ 90 mL/min/1.73m2)
  Interventions: Drug: Evogliptin 5mg

INTERVENTIONS:
Drug: Evogliptin 5mg — Participants receive Single oral administration of Evogliptin 5mg on day1
  Other Names: Suganon
  Arms: Group2
Drug: Evogliptin 5mg — Period 1(1d,After hemodialysis) → Wash-out period → Period 2(15d,Before hemodialysis)
  Hemodialysis patients receive Single oral administration of Evogliptin 5mg on day1 and day15 With a 14-day washout period
  Other Names: Suganon
  Arms: Group1

SUMMARY:
A clinical study to investigate the pharmacokinetics/ pharmacodynamics and safety/tolerability of Evogliptin in hemodialysis patients

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who aged 20 to 80 at the time of screening
2. Subjects with 50.0kg≤Body Weight≤90.0kg and 18.0kg/m2≤BMI≤27.0kg/m2
3. Subjects who meet the following kidney functions

   * group1(hemodialysis patients): MDRD-eGFR ≤ 15 mL/min/1.73m2
   * group2(helthy control): MDRD-eGFR ≥ 90 mL/min/1.73m2

Exclusion Criteria:

1. Subjects who have a uncontrolled or unstable disease such as liver, nervous system, immune system, respiratory system, endocrine system or blood / tumor disease, cardiovascular disease, mental disorders (mood disorder, obsessive compulsive disorder, etc.) or history
2. Subjects who have a gastrointestinal disease (such as Crohn's disease, ulcers, acute or chronic pancreatitis, etc.) or history of gastrointestinal surgery (except simple appendectomy or hernia surgery) that may affect the absorption of the test drug.
3. Subjects with a history of significant hypersensitivity reaction such as anaphylaxis or angioedema to DPP-IV inhibitors
4. Subjects who have AST (SGOT) and ALT (SGPT) greater than 1.5 times the upper limit of normal range, at the time of screening test including additional tests.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

PRIMARY OUTCOMES:
AUClast | 1day(15day) pre-dose (0), 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48 hour post-dose
  Area Under the plasma Concentration versus time curve(AUClast) of Evogliptin
Cmax | 1day(15day) pre-dose (0), 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48 hour post-dose
  Peak Plasma Concentration(Cmax) of Evogliptin

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea